CLINICAL TRIAL: NCT07354165
Title: Assessing Prevalence of Financial Burden and Impact of Cancer on Financial toxicIty in Patients With Early-stage Breast Cancer
Brief Title: Financial Toxicity in Patients With Early-stage Breast Cancer
Acronym: VOICE - GIM36
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: VOICE - GIM36
Record Dates: First submitted 2025-11-25; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: early breast cancer; financial toxicity; quality of life; PROFFIT questionnaire
MeSH Terms: conditions — Breast Neoplasms; Financial Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Cohort 1: patients that received surgery without any further anticancer treatment
  Interventions: Other: Questionnaires
- Cohort 2: patients that received surgery followed by adjuvant chemotherapy only
  Interventions: Other: Questionnaires
- Cohort 3: patients that received surgery followed by chemotherapy and endocrine therapy
  Interventions: Other: Questionnaires
- Cohort 4: patients that received surgery followed by endocrine therapy
  Interventions: Other: Questionnaires
- Cohort 5: patients that received neoadjuvant chemotherapy followed by surgery and no further treatment
  Interventions: Other: Questionnaires
- Cohort 6: patients that received neoadjuvant chemotherapy followed by surgery and adjuvant chemotherapy
  Interventions: Other: Questionnaires
- Cohort 7: patients that received neoadjuvant chemotherapy followed by surgery and adjuvant endocrine therapy
  Interventions: Other: Questionnaires
- Cohort 8: patients that received neoadjuvant endocrine therapy followed by surgery and adjuvant endocrine therapy
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The PROFFIT questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where FT can be expressed and is formed by two type of items: (1) outcome (items 1-7) and (2) determinants (items 8-16). EORTC QLQ-C30, EORTC QLQ-BR42 and HADS questionnaires are currently used in clinical practice

SUMMARY:
Non-profit, multicenter, prospective, observational study. This study aims to evaluate whether the articulated treatment algorithm that is now possible for early-stage breast cancer patients does produce tangible changes of financial distress over the time and whether the determinants of financial distress change their relative weight over the time.

DETAILED DESCRIPTION:
PROFFIT questionnaire is an Italian instrument for evaluating FT in cancer patients in the Italian healthcare context. It includes 16 total items, 7 measuring FT (defining the PROFFIT financial score) and 9 measuring possible determinants of FT. Primary aim of this study is to describe the rate of patients with early breast cancer experiencing financial toxicity (defined as a change of ≥18 points in the PROFFIT-score [items 1-7]) one year after the beginning of the first oncological treatment. In addition, among secondary aims of this study, we aim to verify whether FT is associated with quality of life response , and with disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age > 18 years at the time of study entry
* Histologically confirmed stage I-III invasive breast carcinoma before starting any systemic treatment.

Exclusion Criteria:

* Stage IV invasive breast carcinoma
* Major cognitive dysfunction or psychiatric disorders
* Any previous systemic treatment for the current breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: early-stage breast cancer patients (see cohorts definition)
Sampling Method: Non-Probability Sample
Enrollment: 864 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Financial Toxicity at one year | baseline visit (before surgery or chemotherapy/endocrine therapy depending on the cohort), at the end of chemotherapy/endocrine therapy (if applicable), after surgery, 6 months after surgery, 1 year after the baseline questionnaires
  The rate of patients with early breast cancer experiencing financial toxicity (defined as a change of ≥18 points in the PROFFIT-score [items 1-7]) one year after the beginning of the first oncological treatment

SECONDARY OUTCOMES:
Changes in PROFFIT scores | baseline, at the end of chemotherapy/endocrine therapy (if applicable), after surgery, 6 months after surgery, 1 year after the baseline questionnaires, then every 6 months during endocrine therapy/other treatments/follow-up until 5 yrs from baseline
  baseline PROFFIT-score and its trajectory at subsequent time points across different cohorts and in the whole study sample.
  The Patient Reported Outcome for Fighting FInancial Toxicity (PROFFIT) questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where financial toxicity can be expressed and consist of two type of items: a) outcome (items 1-7) and b) determinants (items 8-16). PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire, range 0-100, 100 indicating maximum financial toxicity.
Financial toxicity "Determinants" | baseline, at the end of chemotherapy/endocrine therapy (if applicable), after surgery, 6 months after surgery, 1 year after the baseline questionnaires, then every 6 months during endocrine therapy/other treatments/follow-up until 5 yrs from baseline
  the individual PROFFIT items (items 8-16 representing potential determinants of financial distress) at baseline and subsequent time points.
  The Patient Reported Outcome for Fighting FInancial Toxicity (PROFFIT) questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where financial toxicity can be expressed and consist of two type of items: a) outcome (items 1-7) and b) determinants (items 8-16). PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire, range 0-100, 100 indicating maximum financial toxicity.
PROFFIT score and survival | baseline, at the end of chemotherapy/endocrine therapy (if applicable), after surgery, 6 months after surgery, 1 year after the baseline questionnaires, then every 6 months during endocrine therapy/other treatments/follow-up until 5 yrs from baseline
  the prognostic role of baseline PROFFIT-score in terms of disease-free survival (DFS), as well as overall survival (OS).
  The Patient Reported Outcome for Fighting FInancial Toxicity (PROFFIT) questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where financial toxicity can be expressed and consist of two type of items: a) outcome (items 1-7) and b) determinants (items 8-16). PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire, range 0-100, 100 indicating maximum financial toxicity.
Quality of Life (EORTC QLQ-C30, EORTC-BR42) | baseline, at the end of chemotherapy/endocrine therapy (if applicable), after surgery, 6 months after surgery, 1 year after the baseline questionnaires, then every 6 months during endocrine therapy/other treatments/follow-up until 5 yrs from baseline
  The prognostic role of baseline PROFFIT-score in terms of QoL outcomes. The Patient Reported Outcome for Fighting FInancial Toxicity (PROFFIT) questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where financial toxicity can be expressed and consist of two type of items: a) outcome (items 1-7) and b) determinants (items 8-16). PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire, range 0-100, 100 indicating maximum financial toxicity.
  EORTC QLQ-C30 scores calculated according to the EORTC QLQ-C30 Scoring Manual; HRQL score calculated by averaging the responses to the items 29 and 30 of the EORTC QLQ-C30; EORTC QLQ-BR42 scores calculated according to the EORTC QLQ-BR42 Scoring Manual.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carmela Piccirillo, MD, Principal Investigator — National Cancer Institute, Naples; Martina Pagliuca, MD, Principal Investigator — Clinical and Translational Oncology, Scuola Superiore Meridionale, Naples
Locations (1):
- National Cancer Institute of Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided